CLINICAL TRIAL: NCT01270360
Title: Validation of a Non Invasive methylateDNA Test for te Diagnosis of Colorectal Tumour in Asymptomatic Individuals
Brief Title: Validation of an Alternative Biological Test to Increase the Detection Sensitivity of a Colon Tumour
Acronym: VATNIMAD
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 09268
Record Dates: First submitted 2010-12-28; First posted 2011-01-05 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Serum Urine, Stools Tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- asymptomatic subjects with positive FOBT: individuals having undergone a positive faecal occult blood test (FOBT) and a reference colonoscopy
  Interventions: Device: COLOHYBRITEST OR VALIHYBRITEST

INTERVENTIONS:
Device: COLOHYBRITEST OR VALIHYBRITEST — Detection of human colon or rectal tumours by using a simplified molecular test based on either a combination of methylated DNA or protein marker(s) alone or considered together in biological fluids like blood, urine and stools

SUMMARY:
Screening campaigns for colorectal cancer (CRC) involve two steps: the detection of occult blood in stools using a Hemoccult GAIAC test (FOBT) on three consecutive stool samples, followed by colonoscopy if the result is positive. The information quality of the Hemoccult test, however, is poor: in the asymptomatic 50 to 74 year-old population, the detection sensitivity of polyps more than 1 cm in diameter is of the order of 10 to 30% and is 35 to 50% for detecting colorectal cancers; specificity is 94 to 98% that of a complete colonoscopy. The I-FOBTs based on immunological detection and quantification of occult blood in stools are currently being evaluated; based on the threshold it can be more sensitive than FOBT, but enhances useless colonoscopies. Alternatively, with highest threshold of blood in stools, it may become highly specific and miss less advanced polyps. Faecal molecular tests based on the detection of human DNA anomalies (point gene mutations, methylation disorders of CG islets) appear to be more sensitive than the detection of occult blood in stools with no loss of specificity, but they are very expensive, thereby limiting their generalisation to the scale of population screening. A formal methylated DNA test has been validated in stools as well as in blood in a cohort of symptomatic individuals having undergone colonoscopy. The aim of the present study is to validate this test by taking advantage of the biotechnical expertise from renowned academic research teams and mass screening organisation.

DETAILED DESCRIPTION:
This study search to validate a test by taking advantage of the biotechnical expertise from renowned academic research teams and mass screening organisation.

In order to reduce the cost of the present study the investigators will select in this preliminary study only those individuals who have a FOBT. However, we'll measure the blood level by using a I-FOBT test to quantify Haemoglobin concentration in stools. Furthermore, we'll use stool DNA to characterize microbiota according to the colonoscopy findings. In addition, the investigators believe it is important to include in the project, the creation of biological blood and urine collections from individuals having undergone both faecal tests and a reference colonoscopy. In the future, these collections will be made available to the national or international scientific community (after consent by the principal investigators) to validate any other molecular and/or protein marker including proteomic analysis by using MSS. The investigators will perform methylated DNA test in either stools or blood and will compare results to those of I-FOBT and colonoscopy.

A simplified molecular test based on a combination of the search for methylation anomalies (one PCR and/or dedicated microarray) a limited number of gene targets involved in colorectal carcinogenesis is available. The investigators will collect stools, urine, and blood in a period of 15 to 2 days prior to colonoscopy. The colonoscopy is performed in 50-74 years old asymptomatic individuals who have presented with a positive FOBT test under mass screening organisation. A final point will be performed 5 years after entry in the trial for all 1000 individuals in order to check occurrence (alternative absence) of any disease during this period and the type of the disease for those individuals who will be shown with normal colonoscopy and to verify evolution of those who will presented with a colon or rectal tumor. Likelihood value of marker in diseases occurring during the survey period will be calculated and prognostic values estimated in those with colon or rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

Every person (actually limited to the average risk of colorectal cancer in national French program):

* having been invited to participate in the organised screening for a colorectal tumour during the study period and having a result positive of the FOBTt
* having given his consent to participate in the study. Patients will be given an information notice at the start of the campaign informing them that participation in this part of the study is optional, to prevent uselessly encumbering the screening campaign operation. Written consent will be obtained before the colonoscopy by the GE for this part of the study
* going to a laboratory to hand over samples of stools, urine and blood prior to the colonoscopy
* being affiliated to social security

Exclusion Criteria:

* Those refusing the colonoscopy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population of asymptomatic subjects selected by a positive faecal occult blood test (FOBT) to undergo colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2010-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine the performances (sensitivity, specificity and likelihood ratios) of a panel of blood and/or faecal molecular DNA markers | 3 years
  To determine the performances (sensitivity, specificity and likelihood ratios) of a panel of blood and/or faecal molecular DNA markers

SECONDARY OUTCOMES:
To estimate the cost and cost-effectiveness of adding DNA molecular tests to FOBT positive patients prior to colonoscopy | 3 years
  To estimate the cost and cost-effectiveness of adding DNA molecular tests to FOBT positive patients prior to colonoscopy
To determine the performances (sensitivity, specificity and likelihood ratios) of a panel of blood and/or faecal molecular protein markers | 3 years
  To determine the performances (sensitivity, specificity and likelihood ratios) of a panel of blood and/or faecal molecular protein markers
To create biological collections for screening purposes (asymptomatic subjects) | 3 years
  To create biological collections for screening purposes (asymptomatic subjects)

CONTACTS AND LOCATIONS:
Overall Officials: Iradj Sobhani, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Derived] Sobhani I, Bergsten E, Charpy C, Chamaillard M, Mestivier D. Virulent Bacteria as Inflammatory and Immune Co-Factor in Colon Carcinogenesis: Evidence From Two Monozygotic Patients and Validation in CRC Patient and Healthy Cohorts. Front Cell Infect Microbiol. 2021 Nov 4;11:749750. doi: 10.3389/fcimb.2021.749750. eCollection 2021. PMID 34804993
- [Derived] Sobhani I, Bergsten E, Couffin S, Amiot A, Nebbad B, Barau C, de'Angelis N, Rabot S, Canoui-Poitrine F, Mestivier D, Pedron T, Khazaie K, Sansonetti PJ. Colorectal cancer-associated microbiota contributes to oncogenic epigenetic signatures. Proc Natl Acad Sci U S A. 2019 Nov 26;116(48):24285-24295. doi: 10.1073/pnas.1912129116. Epub 2019 Nov 11. PMID 31712445